CLINICAL TRIAL: NCT03351881
Title: Nudging Policies in Asia: Evaluating Singapore's Opt-out System for Organ Donation
Brief Title: Evaluation of Attitudes Towards Organ Donation in Individualistic or Collectivistic Countries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSS-1502-P02-02
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Opt Out; Opt In; Opt Neutral

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opt Out (Active Comparator)
  Interventions: Other: Description of Organ Donation Policy
- Opt In (Active Comparator)
  Interventions: Other: Description of Organ Donation Policy
- Opt Neutral (Active Comparator)
  Interventions: Other: Description of Organ Donation Policy

INTERVENTIONS:
Other: Description of Organ Donation Policy — Participants will read about an organ donation policy type (opt-out, opt-in, or opt-neutral) and rate what they think or feel about it.

SUMMARY:
People make decisions every day, both for themselves and on behalf of others. In the case of organ donations, despite the opt-out systems used in Singapore where the default is a presumed consent on the part of the individual, the actualized donation rate is lower than expect. This is partially because family members are called in to make surrogate decisions on behalf of the patient, especially patients near brain death or have been certified to be brain dead.

To address the shortfall in organ donations, the investigators plan to run three studies:

* First, the investigators seek to conduct a representative survey of the public's perception towards organ donation. The investigators will focus on their views towards donating their own vs. family members' organs, and to explore the role of cultural influences on decision-making.
* Second, the investigators will conduct the survey focusing on NUS students and the ways they respond to an opt-out, opt-in, or mandatory organ donation system.
* Third, the investigators will conduct the survey on an online platform (MTurk) to gather the views of participants across India and USA about organ donation.

The studies have the potential to improve actualized organ donation rates, as well as to inform the medical community in their communication with family members.

ELIGIBILITY:
Inclusion Criteria:

* Research participants should be above the age of 21, able to understand English fully, and have no active mental disorder or intellectual impairment.

Exclusion Criteria:

* Below the age of 21, unable to understand English fully, or have active mental disorder or intellectual impairment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Decision to Donate Organ | At the point of the survey, right after participants have read about the organ donation policy condition which they have been assigned.
  Likelihood of participants choosing to donate organs after brain death

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore